CLINICAL TRIAL: NCT01008124
Title: The Liberatory Maneuver for the Treatment of Benign Paroxysmal Positional Vertigo: A Randomized Controlled Trial
Brief Title: The Liberatory Maneuver for the Treatment of Benign Paroxysmal Positional Vertigo (BPPV)
Acronym: LM_BPPV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never recruited/started study
Sponsor: Midwestern University (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Janet Odry Helminski, PhD, Dr, Midwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MWU 1718
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Vertigo; Vestibular Disease
Keywords: Benign Paroxysmal Positional Vertigo; BPPV; PC; BPPN; Vertigo
MeSH Terms: conditions — Vertigo; Vestibular Diseases; Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberatory Maneuver (Experimental): Liberatory Maneuver
  Interventions: Other: Liberatory Maneuver
- Placebo Maneuver (Placebo Comparator): Placebo Maneuver
  Interventions: Other: Placebo maneuver

INTERVENTIONS:
Other: Liberatory Maneuver — 3 cycles of the liberatory maneuver initial session.
  Other Names: Semont Maneuver
  Arms: Liberatory Maneuver
Other: Placebo maneuver — 3 cycles placebo maneuver initial session.
  Arms: Placebo Maneuver

SUMMARY:
This study is being done because the investigators would like to know how effective the Liberatory maneuver is in treating benign paroxysmal positional vertigo (BPPV).

DETAILED DESCRIPTION:
BPPV is a problem with the inner ear that causes brief periods of vertigo triggered by changes in the position of the head such as rolling, looking up, or bending down. BPPV is presently thought to be caused by small pieces of debris or crystals becoming displaced within the inner ear. It can be treated by moving the patient through a series of positions called a maneuver. There are 2 different maneuvers currently used to treat BPPV by the clinician called the liberatory maneuver and the canalith repositioning procedure. We would like to determine how effective the liberatory maneuver is in the treatment of BPPV compared to a placebo maneuver.

ELIGIBILITY:
Inclusion Criteria:

* BPPV involving the posterior canal on only one side

Exclusion Criteria:

* No other canals involved (anterior canal or lateral canal), no central nervous system disorder, and no other medical condition that would not enable the individual to have the maneuver done.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11 (Estimated); Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Negative Dix-Hallpike maneuver | 1-2 weeks

SECONDARY OUTCOMES:
Self reported willingness to move | 1-2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janet O. Helminski, PhD, Principal Investigator — Midwestern University
Locations (2):
- United States (2):
  - Chicago Dizziness and Hearing, Chicago, Illinois
  - Midwestern University, Downers Grove, Illinois

REFERENCES:
- [Background] Salvinelli F, Trivelli M, Casale M, Firrisi L, Di Peco V, D'Ascanio L, Greco F, Miele A, Petitti T, Bernabei R. Treatment of benign positional vertigo in the elderly: a randomized trial. Laryngoscope. 2004 May;114(5):827-31. doi: 10.1097/00005537-200405000-00007. PMID 15126738
- [Background] Massoud EA, Ireland DJ. Post-treatment instructions in the nonsurgical management of benign paroxysmal positional vertigo. J Otolaryngol. 1996 Apr;25(2):121-5. PMID 8683652